CLINICAL TRIAL: NCT00005506
Title: Vascular Disease--Structure/Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5024; R01HL059503 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To investigate the relationship of non-invasively measured flow-mediated brachial artery dilation with coronary artery disease (CAD).

DETAILED DESCRIPTION:
BACKGROUND:

This study meshed with a longitudinal case-control study, HL-35333, Carotid Atherosclerosis Follow-Up Study. HL-35333 comprised 280 individuals older than 45 equally divided between men and women, half with and half without CAD evaluated for risk factors at baseline and with completed follow-up with yearly B-mode for three years. The Carotid Atherosclerosis Follow-Up Study quantified the interassociations of angiographically defined coronary artery disease and CAD risk factors with progression. The NIH funded a continuation of this effort to review existing ultrasound tapes from this study in order to additionally evaluate the associations of all these factors with extracranial carotid arterial dimensions (ECAD: interadventitial and lumen diameters) and change in ECAD over time.

DESIGN NARRATIVE:

The study assessed brachial artery reactivity among 100 CAD subjects and 100 controls who had been previously enrolled in a study of the relationship between extracranial intima media thickness (ECIMT) as assessed by B mode ultrasonographic measurements and CAD status. Most subjects had three consecutive B mode measurements at 12 month intervals. These subjects had brachial artery reactivity measurements according to a standardized protocol. Linear regression analysis was used to relate brachial artery reactivity to CAD status, gender and risk factors as predictors. Interaction effects were also assessed between CAD status and other risk factors and also between gender and other risk factors. Similar analyses were performed to relate percent dilation to ECIMT measurements.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Crouse, III — Wake Forest University

REFERENCES:
- [Background] Espeland MA, Tang R, Terry JG, Davis DH, Mercuri M, Crouse JR 3rd. Associations of risk factors with segment-specific intimal-medial thickness of the extracranial carotid artery. Stroke. 1999 May;30(5):1047-55. doi: 10.1161/01.str.30.5.1047. PMID 10229743
- [Background] Herrington DM, Fan L, Drum M, Riley WA, Pusser BE, Crouse JR, Burke GL, McBurnie MA, Morgan TM, Espeland MA. Brachial flow-mediated vasodilator responses in population-based research: methods, reproducibility and effects of age, gender and baseline diameter. J Cardiovasc Risk. 2001 Oct;8(5):319-28. doi: 10.1177/174182670100800512. PMID 11702039
- [Background] Terry JG, Tang R, Espeland MA, Davis DH, Vieira JL, Mercuri MF, Crouse JR 3rd. Carotid arterial structure in patients with documented coronary artery disease and disease-free control subjects. Circulation. 2003 Mar 4;107(8):1146-51. doi: 10.1161/01.cir.0000051461.92839.f7. PMID 12615793